CLINICAL TRIAL: NCT04536636
Title: Effect of Oral Administration of Docohexanoic Acid on Anemia-inflammation in Hemodialysis Patients. A Randomized Clinical Trial
Brief Title: Docohexanoic Acid in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHA-HD (188-16)
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The patients on this arm received usual medical care
  Interventions: Drug: Control-No drug
- DHA supplementation (Active Comparator): The patients on this arm received DHA supplementation (650 mg DHA/3 times/wk/post-HD session)
  Interventions: Drug: Docohexanoic acid

INTERVENTIONS:
Drug: Docohexanoic acid — Patients received 650 mg DHA/3 times/wk/post-HD session
  Arms: DHA supplementation
Drug: Control-No drug — Patients received usual medical care with no DHA
  Arms: Control

SUMMARY:
Docohexanoic acid (DHA), a dietary n-3 polyunsaturated fatty-acid omega-3 (n-3, PUFA), showed potential beneficial effects in reducing all-cause mortality in hemodialysis (HD) patients. This clinical trial aimed to analyze whether DHA supplementation was a modulator of erythropoietin (EPO) response and inflammation in hemodialysis (HD) patients.

DETAILED DESCRIPTION:
Background. Docohexanoic acid (DHA), a dietary n-3 polyunsaturated fatty-acid omega-3 (n-3, PUFA), showed potential beneficial effects in reducing all-cause mortality in hemodialysis (HD) patients. This clinical trial aimed to analyze whether DHA supplementation was a modulator of erythropoietin (EPO) response and inflammation in hemodialysis (HD) patients.

Methods. In single-blind, controlled clinical trial, 52 HD patients were randomized to either DHA supplementation (650 mg DHA/3 times/wk/post-HD session) or controls (usual medical-care) for 8-weeks. Clinical data by collecting hemoglobin concentration (Hb), weekly dose of EPO, and erythropoietin resistance index (ERI). The inflammatory response was measured using serum C-reactive protein (s-CRP) and plasma homocysteine (tHcy) at baseline (T0) and post-intervention (T1). miR-146a array was used as an inflammatory biomarker. Post-intervention measures were analyzed at 4-weeks intervals and adjusted by baseline in a linear regression.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* chronic stabilized HD treatment for at least 3 months with functional vascular access (arteriovenous fistula or permanent catheter)
* equilibrated Kt/V urea (eKt/V)higher than 1.2
* informed consent form signed

Exclusion Criteria:

* exposure to corticosteroids and anti-inflammatory drugs or hospital admissions in last 3 months
* were with ongoing active illnesses, wasting, connective tissue disease, metastatic cancer or malignancy, HIV, uncontrolled chronic hepatic disease or transplantation prior to the start of the study.
* Patients with known hypersensitivity to any of fish intolerance or allergy, history of gastrointestinal bleeding, patients already receiving chronic anticoagulation therapy (antiplatelet agents or warfarin), and patients with terminal or life-threatening disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Determine correction of anemia | Determine correction of anemia measured by erythropoiesis-resistance index (ERI) to detect a difference of 10 units of response between groups at 8 weeks follow-up, with a SD of 10 and a power higher than 80%.
  Determine correction of anemia measured by erythropoiesis-resistance index (ERI) to detect a difference of 10 units of response between groups at 8 weeks follow-up, with a SD of 10 and a power higher than 80%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Derived] Ruperto M, Rodriguez-Mendiola N, Diaz-Dominguez M, Gimenez-Moyano S, Garcia-Bermejo ML, Fernandez-Lucas M. Effect of oral administration of docohexanoic acid on anemia and inflammation in hemodialysis patients: A randomized controlled clinical trial. Clin Nutr ESPEN. 2021 Feb;41:129-135. doi: 10.1016/j.clnesp.2020.12.004. Epub 2020 Dec 31. PMID 33487255